CLINICAL TRIAL: NCT06714058
Title: Cardiometabolic Risk of Obese Subjects: Cross-sectional Study for the Identification of Genetic, Laboratory and Clinical Determinants
Brief Title: Cardiometabolic Risk of Obese Subjects: Cross-sectional Study
Acronym: MiRNome
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MiRNome
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Obesity-related Medical Conditions; Cardiovascular Risk; Genetics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — study-specific blood sampling for the evaluation of the expression profile of circulating miRNAs, the search for variants of the HMGA1 gene and the assay of the HMGA1 protein, of circulating biomarkers of inflammation and insulin resistance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
experimental study with analysis on tissues. This study aims to study cardiometabolic risk from a genetic, clinical, instrumental and laboratory point of view in a population of subjects with obesity.

DETAILED DESCRIPTION:
Compared to normal clinical practice, if you decide to participate in the study you will be asked to:

1. allow the collection of an additional study-specific amount of blood as part of a blood sample already provided for by clinical practice during the dietetic visit; The sample will be used to perform the genetic and laboratory analyses required by the study.
2. Undergo an additional study-specific visit within one month of the dietetic visit. will be subjected to the measurement of the degree of vascular aging and the evaluation of the health of his/her arteries, through non-invasive examinations.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years

  * BMI > 30 Kg/m2
  * In primary prevention for cardiovascular disease
  * Ability to communicate, make themselves understood and adhere to study-specific procedures
  * Willingness to participate in the study and obtain informed consent

Exclusion Criteria:

* Patients already enrolled by the Research Units involved in the enrolment
* Glycated hemoglobin level > 55 mmol/L
* Patients suffering from obesity secondary to endocrinological diseases or iatrogenic causes
* Patients with heterozygous Familial Hypercholesterolemia (Dutch Lipid Score - DLS>8)
* Patients suffering from hypercholesterolemia secondary to lipid or iatrogenic extra-metabolic pathologies
* Patients suffering from systemic inflammatory or oncological diseases
* Patients on active treatment with GLP-1 analogues
* Pregnancy and breastfeeding
* Any medical or surgical condition that makes the patient's adherence to the study protocol complex or inconsistent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients of both sexes, suffering from grade I obesity, not suffering from atheromatous cardiovascular diseases (ischemic heart disease, ischemic stroke, peripheral arterial disease)
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
cycle threshold miRNAs | at baseline
  Study of the expression profile of specific circulating miRNAs
Presence/absence of the loss-of-function HMGA1 allelic variant (rs146052672) | baseline
  search for variants of the HMGA1 gene
NGS sequencing of the genes: MC4R, LEP, LEPR, POMC, PCSK1, ADRA2, AGPAT2, HIF1A, HMGA2, HMGB1, INSR, PEPCK, GLUT/SGLT glucose transporters. | baseline
  NGS expression of the genes: MC4R, LEP, LEPR, POMC, PCSK1, ADRA2, AGPAT2, HIF1A, HMGA2, HMGB1, INSR, PEPCK, GLUT/SGLT glucose transporters.
Insulinemia (µU/mL) | baseline
  Levels of haematic insulin
C-peptide (nmol/L) | baseline
  Levels of haematic of C-peptide
thyrotropin (nmol/L) | baseline
  Levels of haematic of thyrotropin
HMGA1 protein assay | baseline
  Levels of haematic HMGA1 protein

CONTACTS AND LOCATIONS:
Overall Officials: Maria Letizia Petroni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - Maria Letizia Petroni, Bologna, BO
  - Azienda Ospedaliero-Universitaria "Renato Dulbecco" di Catanzaro, Catanzaro